CLINICAL TRIAL: NCT05948904
Title: Defining a Technique for the Use of Cryogenic Catheters for Biopsy and Ablation for the Diagnostic and Treatment of Pulmonary Lesions: An Ex-Vivo Human Lung Model Study.
Acronym: CT0129
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-11550
Record Dates: First submitted 2023-05-23; First posted 2023-07-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Lung Diseases
Keywords: Lung; cryobiopsy; cryoablation; transbronchial intervention
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ex Vivo Cryo (Experimental): Multiple procedures will be performed to each model in order to accomplish the objectives of the study. Tissue samples will be taken from the models and images will be performed. This will allow us to determine which configuration is the optimal for obtaining the more effective and stable models that could offer the best quality specimens as well.
  Interventions: Diagnostic Test: Cryo Ex Vivo

INTERVENTIONS:
Diagnostic Test: Cryo Ex Vivo — Lungs from patients undergoing lung transplantation after their removal from the recipient patient with previous informed consent signed before transplantation will be obtained. The organs will be placed in an acrylic box and will be kept at a temperature of 37 Celsius degrees. The lungs will be mechanically ventilated connected by an endotracheal tube size 8 inserted in the bronchus with the balloon inflated and a silk suture providing a hermetic closure proximal to the balloon.
  Tissue samples will be taken from the models and images will be performed.

SUMMARY:
Developing a standardized methodology for the use of novel cryogenic catheters for transbronchial cryobiopsy and cryoablation of pulmonary lesions.

DETAILED DESCRIPTION:
Surgical lung biopsy (SLB) and surgical resection are the current gold standard for both tissue sampling and ablation of pulmonary lesions. Albeit the use of minimally invasive surgical techniques (VATS), these interventions are frequently associated with complications which include: prolonged air leak, pneumonia, prolonged length of stay in the intensive care unit as well as an increased mortality rate which is influenced by the nature (elective vs non-elective) of the case. To reduce trauma to patients, transbronchial interventions are becoming increasingly popular. However, current techniques have only been demonstrated in humans for lung biopsy and often provide lesser quality specimens than SLB. Promising results have been achieved using cryotechnology but a standardized technique has yet to be established.

To demonstrate the potential for transbronchial interventions using cryo, we aim to develop a standardized technique for transbronchial cryobiopsy and cryoablation of pulmonary lesions using a human ex-vivo model.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lung transplant surgery

Exclusion Criteria:

* Organ donor ineligible to donate lungs
* Healthy individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Measure of Pleural breakage (Absent or Present) | 48 months
  Develop a standardized methodology for the use of novel cryoprobes for transbronchial lung biopsies and ablation of pulmonary lesions
Temperature of ice ball at center; Temperature of ice ball at periphery; Temperature of ice ball at varying distances from ice ball | 48 months
  Develop a standardized methodology for the use of novel cryoprobes for transbronchial lung biopsies and ablation of pulmonary lesions
Model of cryogen | 48 months
  Develop a standardized methodology for the use of novel cryoprobes for transbronchial lung biopsies and ablation of pulmonary lesions
Freezing Time | 48 months
  Develop a standardized methodology for the use of novel cryoprobes for transbronchial lung biopsies and ablation of pulmonary lesions
Size of resected specimen | 48 months
  Develop a standardized methodology for the use of novel cryoprobes for transbronchial lung biopsies and ablation of pulmonary lesions

SECONDARY OUTCOMES:
Blood loss and complication | 48 months
  Feasibility of transbronchial lung cryobiopsy and cryoablation

CONTACTS AND LOCATIONS:
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No